CLINICAL TRIAL: NCT05692726
Title: Evaluation of Volume and Electrolyte Balance in Hyponatremia Treatment - a Prospective Observational Trial (EvenT)
Brief Title: Evaluation of Volume and Electrolyte Balance in Hyponatremia Treatment - a Prospective Observational Trial
Acronym: EvenT
Status: Recruiting | Type: Observational
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Volker Burst, Prof. Dr., University of Cologne
Other Study IDs: V1.0-20220315
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Non-hypervolemic Hyponatremia
Keywords: Electrolyte-free water clearance; hyponatremia
MeSH Terms: conditions — Hyponatremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients with non-hypervolemic hypotonic hyponatremia
  Interventions: Other: Patients

INTERVENTIONS:
Other: Patients — Patients will get study-specific measurements within first 5 days of standard of care treatment of hyponatremia or until discharge

SUMMARY:
To assess quantitatively the evolution over time of electrolyte-free water clearance and electrolyte mass balance in patients with non-hypervolemic hypotonic hyponatremia

DETAILED DESCRIPTION:
Achieving recommended treatment targets in management of hyponatremia is challenging: plasma sodium must be increased effectively but, at the same time, overcorrection has to be prevented. Yet, predictors of change of sodium over time have not been delineated properly. It was found, that evidence hinting to the fact that sodium baseline itself is crucial with respect to sodium evolution.

The goal of this study is to gather prospective data in order to precisely delineate the role of initial sodium levels by correlating those to plasma sodium evolution and electrolyte free water evolution. It is aimed to decipher patterns of sodium evolution with respect to anthropometric data, such as body composition analyses and blood pressure and markers of innate regulation mechanisms of body volume like aldosterone and renin. In addition, apart from these clinical aspects, a better appreciation of the physiological responses to hyponatremia treatment in terms of water and electrolyte balances is undoubtedly necessary to improve understanding of the body's mechanisms involved in osmotic homeostasis and cell volume control. Since studies to date also lack consideration of the intracellular department, the aim is to close that gap.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years
* Hypotonic hyponatremia

  * glucose-corrected plasma sodium <130 mmol/l
  * serum osmolality <280 mosmol/kg or lack of signs of non-hypotonic hyponatremia

Exclusion Criteria:

* Signs of extracellular volume expansion
* Patients with liver cirrhosis and severe liver damage AST/ALT>3xULN, AP>6xULN, Bilirubin ≥ 3mg/dl
* Patients with heart failure
* Patients on dialysis and/or patients with oliguric renal impairment and plasma creatinine ≥ 3mg/dl
* Patients after organ transplantation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with non-hypervolemic hyponatremia
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-10-15 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Plasma Sodium | baseline, every day up to 30 days
  Measurement of plasma sodium in blood samples
Changes in plasma osmolality | baseline, every day up to 30 days
  Measurement of plasma osmolality for determination of electrolyte-free water clearance before, during and after hyponatremia treatment
Changes in urine osmolality | baseline, every day up to 30 days
  Determination of electrolyte-free water clearance before, during and after hyponatremia treatment by measurement of urine osmolality
Changes in urine volume | baseline, every day up to 30 days
  Determination of electrolyte-free water clearance before, during and after hyponatremia treatment by measurement of urine volume

SECONDARY OUTCOMES:
Changes in body weight | baseline, every day up to 30 days
  Measurement of body weight before, during and after hyponatremia treatment by bioimpedance measurement
Changes in total body water | baseline, every day up to 30 days
  Measurement of body water before, during and after hyponatremia treatment by bioimpedance measurement
Changes in intracellular volume | baseline, every day up to 30 days
  Measurement of intracellular volume before, during and after hyponatremia treatment by bioimpedance measurement
Changes in extracellular volume | baseline, every day up to 30 days
  Measurement of extracellular volume before, during and after hyponatremia treatment by bioimpedance measurement
Changes in blood pressure | baseline, every day up to 30 days
  Measurement of blood pressure before, during and after hyponatremia treatment
Changes in cell size | baseline, every day up to 30 days
  Determination of blood cell size via measurement of mean corpuscular volume
Changes in intracellular electrolyte levels | baseline, every day up to 30 days
  Measurement of whole blood samples via ICP-mass spectrometry
Changes in copeptin levels | baseline, every day up to 30 days
  Measurement of copeptin in blood samples
Changes in renin levels | baseline, every day up to 30 days
  Measurement of renin in blood samples
Changes in aldosterone levels | baseline, every day up to 30 days
  Measurement of aldosterone in blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Volker Burst, MD, Prof., Principal Investigator — University Hospital of Cologne
Locations (1):
- University Hospital of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No